CLINICAL TRIAL: NCT04503811
Title: Exploring the Lived Experience of Control and Wellbeing of Older Persons Diagnosed With Frailty Within the Care Service Provision in Southern England
Brief Title: Sense of Control in Frail Older Persons
Acronym: CONtrol
Status: Completed | Type: Observational
Sponsor: Bournemouth University (Other)
Responsible Party: Sponsor
Other Study IDs: AN282540
Record Dates: First submitted 2020-08-05; First posted 2020-08-07 (Actual); Last update posted 2022-03-02 (Actual); Status verified 2022-03

CONDITIONS: Frailty; Older People; Sense of Control
MeSH Terms: conditions — Frailty

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Other
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Frail Older People: The first phase of the data collection process will include one to one interviews with up to twenty (20) frail older people. The pre-selected inclusion criteria for this category of participants include; older people (aged 65 years and over); individuals diagnosed with frailty and receiving (part of their) care services at the Day Hospital; the capacity to give free and fully informed consent; ability to use the English language, as well as judgement by the clinical staff and/or nominated manager that the potential participant can take part in an in-depth interview.
- Day Hospital Staff: The second phase of the data collection process will entail one to one interviews with up to ten (10) Staff at the Day Hospital. The study will include staff that routinely work with frail older people at the Day Hospital including nurses (registered and unregistered), doctors, physiotherapists, occupational therapists and therapy assistants that can give free and fully informed consent. Furthermore, the study will include both part-time and full-time staff with a minimum of six months of work experience with frail older people.

SUMMARY:
The proposed study seeks to explore the lived experience of control and wellbeing of older people diagnosed with frailty within the care service provision in southern England.

In the study, the researcher will talk with older people diagnosed with frailty and the professionals that provide care to them. The researcher is interested in understanding participants' experiences of a sense of control and how health and social care services affect this experience.

Although research has shown that rehabilitation can be effective in maintaining physical activity often frail older people do not wish to take up the rehabilitation services provided. Research in this area has been dominated by health care professionals' views about frailty and how services should be provided. Services could be improved by learning from the first-hand experiences of older people living with frailty and what they feel increases their level of control and wellbeing within their service use. The factors which increase their sense of control and wellbeing can then be built into future service development, inform care policies, and provide new understanding for future research to develop services which are more attractive and relevant for older frail people.

All persons aged 65 years and over, with a diagnosis of frailty will be eligible to take part in one to one interviews with the researcher. From the interviews principles underpinning good practice which enhances the sense of control and wellbeing in older people's lives and within the services received will be identified. These will be shared with professional care providers including nurses, doctors, and physiotherapists who routinely work with frail older people to gain insights into how these principles can be integrated into practice and developed in policy and future service development. The findings will, therefore, help to develop services which ensure that they are supportive and increase a sense of control in life rather than getting in the way of this.

The study is expected to last 12 months and up to 30 participants (20 older people and 10 Hospital staff) will be recruited to take part in the study.

ELIGIBILITY:
Inclusion Criteria:

Phase one inclusion criteria (frail older people) The pre-selected inclusion criteria for this category of participants include;

* older people (aged 65 years and over);
* individuals diagnosed with frailty and receiving (part of their) care services at the Day Hospital;
* the capacity to give free and fully informed consent;
* ability to use the English language, as well as judgement by the clinical staff and/or nominated manager that the potential participant can take part in an in-depth interview.

Phase two inclusion criteria (Hospital staff)

* The study will include staff that routinely work with frail older people at the Day Hospital including nurses (registered and unregistered), doctors, physiotherapists, occupational therapists and therapy assistants that can give free and fully informed consent.
* Furthermore, the study will include both part-time and full-time staff with a minimum of six months of work experience with frail older people.

Exclusion Criteria:

Phase one exclusion criteria

The exclusion criteria, on the other hand, will include:

* people who cannot communicate in English;
* and individuals who are acutely medically unwell.

Phase two exclusion criteria

The second phase of the study will, on the other hand, exclude:

• all staff who do not have routine direct contact with patients' care, for example, the senior managers.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: The study will focus on frail older people and Day Hospital staff that provide care to them.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2021-09-15 (Actual); Primary Completion 2022-02-21 (Actual); Study Completion 2022-02-21 (Actual)

PRIMARY OUTCOMES:
How frail older people understand and experience control in their lives and care | Up to one and a half hours
  The study will highlight frail older people's experiences, opinions and viewpoints on their sense of control in their lives and care processes and how this impacts on their dignity and well-being.
How frail older peoples' experiences can be used to shape and enhance care design and delivery. | Up to one and a half hours
  The study will aslo highlight how health and social care practices can draw from older people's experiences to inform the design and delivery of care services.
How professional care providers can integrate into care practice principles that enhance service users' sense of control and well-being. | Up to one hour
  The study will help professional care providers working with older people to develop services which ensure that they are supportive and increase a sense of control in life rather than getting in the way of this.

CONTACTS AND LOCATIONS:
Overall Officials: Caroline Ellis-Hill, Study Director — Chief Investigator/Senior Lecturer In Qualitative Research
Locations (1):
- University Hospitals Dorset NHS Foundation Trust, Bournemouth, Christchurch, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
The researcher will ensure that the Data is made open and accessible to other researchers in line with the provisions of the InnovateDignity Project Data Management Plan and the Bournemouth University Research Data Policy.
  Once the study has ended, anonymised data from the project will be deposited in the 'UK Data Archive' in Qualibank for example and QuDEX as a way of ensuring that the data are easily accessible to other researchers in the specific field of study and/or social scientists in related fields such as health care and policy research. However, there will be an embargo of up to 3 years on publications, after which data will be made available and accessible via the UK Data Archive.
  The data will be secured in line with the UK Data Archive policies and at the end of the project and the three-year embargo, researchers seeking access to the data will have to go through the UK Data Service access processes.
Supporting Information: Study Protocol
Time Frame: The data will become available three years after the end of the project.
Access Criteria: The data will be secured in line with the UK Data Archive policies and at the end of the project and the three-year embargo, researchers seeking access to the data will have to go through the UK Data Service access processes.
URL: http://ukdataservice.ac.uk/